CLINICAL TRIAL: NCT02819128
Title: Investigation of Endemic and Emerging Diseases in Populations of Homeless Households in Marseille.
Acronym: SDF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-44
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Endemic and Emerging Diseases in Populations of Homeless
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Homeless people (Other): Populations of homeless households in Marseille.
  Interventions: Other: Swabs skin, pharyngeal, and blood sample; Other: Collection of body lice

INTERVENTIONS:
Other: Swabs skin, pharyngeal, and blood sample — Collection of one blood sample with a volume of 10 mL (2 tubes of blood 5 mL ) and 2 swabs ( throat and skin ).
Other: Collection of body lice — For the subjects infested with body lice , if they want, their underwear will be recovered and sent to the laboratory to measure the resistance to permethrin.

SUMMARY:
Hypothesis:

Homeless people have infections not diagnosed with a potential impact on their health status.

Main Purpose: Improve the etiological diagnosis of endemic and/or emerging pathologies among homeless people.

DETAILED DESCRIPTION:
In Marseilles, the population of homeless is estimated at 1500 individuals, including 800 usually sleeping in the street, 600 in foster homes and a hundred in the structures of care. The precarious living conditions of homeless persons promote the emergence or re-emergence of many communicable infectious diseases homeless people whose symptoms are often overlooked by the subject and rarely established etiologic diagnosis.

Among these diseases, frequently described in the literature are infestation by lice and infectious diseases that they transmit (Bartonella quintana), skin infections, hepatitis E and C and finally the infection with Tropheryma Whipplei. In this study we propose to systematically in homeless subject an etiological diagnosis of pathogens at the origin of these diseases (i) to improve knowledge (ii) to improve their management, (iii) to limit the contagion.

ELIGIBILITY:
Inclusion Criteria:

* Homeless Subject on the day of the study in one of two shelters for homeless Marseille ( Madrague City and Forbin )
* Major subject ( > or equal to 18 years)
* Freely about having signed the written informed consent,
* About affiliated with a social security scheme

Exclusion Criteria:

* Minor Subjects ( < 18 years )
* Major subject under guardianship (L. 1121-8 )
* Subject privated of freedom or under court order (L. 1121-6 )
* Subject refusing to sign the informed consent form ,
* Subject not affiliated with a social security insurance
* Pregnant women , parturient or nursing (L. 1121-7 ) .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2014-01-25 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with an established microbiological diagnosis | 3 years

SECONDARY OUTCOMES:
Prevalence of skin infections | 1 day
Prevalence of Tropheryma whipplei infections | 1 day
Prevalence of infestation by body lice | 1 day
Percentage of body lice resistant to permethrin | 1 day
Prevalence of infections by Bartonella quintana | 1 day
Prevalence of infection by hepatitis E and C | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BROUQUI, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided